CLINICAL TRIAL: NCT01123213
Title: Characteristics Predictive of Pessary Success
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Karen Noblett, Division Director, University of California, Irvine
Other Study IDs: 2008-6704
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: All Patients Who Have Undergone a Pessary Fitting
Keywords: pelvic organ prolapse; pessary fitting
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pessaries are mechanical support devices worn vaginally to treat the symptoms of pelvic organ prolapse, such as vaginal pressure or a vaginal bulge. Pessaries are one of the options along with surgery and expectant management for pelvic organ prolapse. As the aging population grows, more patients will need treatment for pelvic organ prolapse. Various studies have been conducted previously to identify patient parameters predictive of successful pessary fitting and continued use. Our study is a retrospective chart review to identify patient characteristics predictive of successful pessary fitting and use, specifically focusing on the parameters of POPQ, pelvic organ prolapse quantification exam, and the ratio of the genital hiatus, which is the length of the vaginal opening, and total vaginal length.

ELIGIBILITY:
Inclusion Criteria:

* undergone a pessary fitting by physicians in the division of Urogynecology between the years of 2000 to 20008.

Exclusion Criteria:

* Patients will be excluded only if their chart does not contain the clinical data under review.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone a pessary fitting by physicians in the division of Urogynecology between the years of 2000 to 20008 will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — UCI Medical Center
Locations (1):
- UC Irvine Women's Healthcare, Orange, California, United States